CLINICAL TRIAL: NCT04100369
Title: Admission Blood Glucose as a Predictor of Morbidity and Mortality in Polytraumatized Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, tamer refaat hanna armanious, Assistant Lecturer, Assiut University
Other Study IDs: blood glucose
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Blood Glucose, High
Keywords: shock , poly trauma , serum lactate
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laboratory — Arm

SUMMARY:
In polytrraumatized patients, Does hyperglycaemia on admission increase the risk of morbidity and mortality compared to polytraumatised patients with normal blood glucose level ?

DETAILED DESCRIPTION:
Trauma is still the leading cause of death in young adults and a major cause of morbidity and mortality at all ages.(1,2). Polytrauma is defined as injury to several physical regions or organ systems, where at least one injury or the combination of several injuries are life threatening with the severity of injury being equal or >16 on the scale of the Injury Severity Score (ISS). Prediction of mortality in trauma patients is an important part of trauma care (3). The trauma and injury severity score (TRISS) and Acute Physiology and Chronic Health Evaluation IV (APACHE IV) are used commonly to predict injury severity and risk of mortality. Although it is regarded as the international standard in trauma scoring, it has complex calculating and incorporates the Glasgow Coma Scale (GCS) for neurological evaluation (4). Regardless of the accuracy of trauma scores, is based on an anatomical description of every injury and cannot be assigned to the patients until a full diagnostic procedure has been performed(5) . Many studies have revealed alteration in glucose metabolism in trauma and proportional relation of its high level to the degree of injury (6). hyperglycaemia is associated with similar complications as uncontrolled diabetes, including an increased mortality, an increased number of infectious complications, and poor wound healing. The presence of elevated blood glucose also impedes normal host defences against infection and impairs the normal inflammatory response (7.8).

* Therefore, this study will be conducted to compare between alterations in easy and rapid predictors as glucose level, base deficit and lactate and difficult and slow predictors as TRISS and APACHE IV. So, it could be considered an early and easy rapid predictor of outcome .

ELIGIBILITY:
Inclusion Criteria:

* • Age >= 18 years

  * Polytrauma ISS >= 18
  * Recent polytrauma patients who are directly transferred by the ambulance from the scene of accident to assiut university hospital and did not receive resuscitative measurements in another hospital

Exclusion Criteria:

* known co-morbidities affecting blood glucose level like :

  * Pregnant women
  * Diabetic patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: using blood glucose as an easy and a rapid predictor of morbidity and mortality in poly traumatized patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Admission blood glucose as a predictor of morbidity and mortality in polytraumatized patients | baseline
  to investigate the admission blood glucose level as a predictor of morbidity and mortality in poly traumatized patients

SECONDARY OUTCOMES:
Admission blood glucose as a predictor of morbidity and mortality in polytraumatized patients | baseline
  correlation of blood glucose level to serum lactate , interlukin6 , C reactive protein , coagulation profile and their use as biomarkers in polytraumatized patients

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Abubeih, ass.prof, Study Director — Assiut University; fasil adam, prof, Study Director — Assiut University

REFERENCES:
- [Background] Laird AM, Miller PR, Kilgo PD, Meredith JW, Chang MC. Relationship of early hyperglycemia to mortality in trauma patients. J Trauma. 2004 May;56(5):1058-62. doi: 10.1097/01.ta.0000123267.39011.9f. PMID 15179246
- [Background] Lichtveld RA, Panhuizen IF, Smit RB, Holtslag HR, van der Werken C. Predictors of Death in Trauma Patients who are Alive on Arrival at Hospital. Eur J Trauma Emerg Surg. 2007 Feb;33(1):46-51. doi: 10.1007/s00068-007-6097-6. Epub 2007 Feb 27. PMID 26815974